CLINICAL TRIAL: NCT03368482
Title: Brain Gym® Exercises for Institutionalized Elderly People With Cognitive Impairment: Findings From a Comparative Study.
Brief Title: Brain Gym® Exercises for Institutionalized Elderly People With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, José M. Cancela, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-2402-16
Record Dates: First submitted 2017-11-28; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Cognition Disorders in Old Age; Physical Activity
Keywords: cognition disorders; frail elderly; human physical conditioning; institutionalization; physical activity
MeSH Terms: conditions — Motor Activity; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain Gym Exercises (Experimental): Brain Gym® (BG) is a movement-based program originally designed to improve learning capabilities through the performance of mind-body exercises. BG can be considered as an interesting field of research due to the need of identifying novel therapies which might be more pleasant for older adults who tend not to be prone to participating in conventional exercise programs and might have a positive effect on their cognitive function. In spite of this, scientific evidence regarding the effects of BG on people with cognitive impairment is scarce.
  Interventions: Behavioral: Brain Gym Exercises
- Standard Exercises (Active Comparator): A traditional physical exercise program designed for institutionalized elderly people aimed at increasing their range of mobility and coordination, specifically focused on the lower limbs.
  Interventions: Behavioral: Standard exercise program for institutionalized older adults.

INTERVENTIONS:
Behavioral: Brain Gym Exercises — Participants in the BrainGym Exercises group performed six of the following BG exercises in every training session they took part in: "Cross Crawl", "Gravity Glider", "Arm Activation", "Belly Breathing", "Hook-ups", "Think of an X", "Lazy Eights", "Elephant", "Space Buttons", "The Owl", "Energy Yawn", "Balance Buttons" and "The Energizer". All exercises were executed from a sitting position but following the main tenets of the Brain Gym® work routine.
  Arms: Brain Gym Exercises
Behavioral: Standard exercise program for institutionalized older adults. — Participants in the Standard Exercise group took part in a traditional physical exercise program designed for institutionalized elderly people aimed at increasing their range of mobility and coordination, specifically focused on the lower limbs.
  Arms: Standard Exercises

SUMMARY:
Scientific evidence regarding the effects of Brain Gym®, on people with cognitive impairment is scarce. This study aimed at comparing the effects of a program based on Brain Gym® exercises against a fitness exercise program on the cognitive function, functional independence, physical fitness and quality of life in institutionalized older adults with cognitive impairment.

DETAILED DESCRIPTION:
Cognitive training and physical exercise have been regarded as useful strategies in order to improve the cognitive function in older people with cognitive impairment. In this regard, it has been argued that while physical exercise improves the metabolic activity of the brain, the performance of cognitively demanding tasks increases the amount of dendritic branches and the level of synaptic plasticity, implying that the combination of both therapies may result in synergistic effects that positively influence various cognitive domains in different ways. One of the best known therapies which combines mental and physical training is Brain Gym® (BG), a movement-based program originally designed to improve learning capabilities through the performance of mind-body exercises. Brain Gym® can be considered as an interesting field of research due to the need of identifying novel therapies which might be more pleasant for older adults who tend not to be prone to participating in conventional exercise programs and might have a positive effect on their cognitive function. In spite of this, scientific evidence regarding the effects of BG on people with cognitive impairment is scarce and none of the studies compared the potential benefits of BG versus traditional exercise programs for this population. Moreover, to the authors' knowledge no study of this kind has been published so far. Under these circumstances, the present study aims at identifying the potential benefits of performing BG exercises on the cognitive function, functional independence, physical fitness, and quality of life of institutionalized older people with cognitive impairment, as well as at finding out whether the effects are more significant than those produced by a traditional exercise program.

ELIGIBILITY:
Inclusion criteria:

* Older than 65 years old.
* Mean score ≤ 24 in the Spanish adapted version of the Mini-Mental State Examination.
* Cognitive and co-operative ability to follow simple instructions.

Exclusion criteria:

• Individuals whose medical condition hindered or prevented their full and complete participation in the evaluation tests.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Assessment of the changes in participants' cognitive function. | 10 weeks
  By means of the Spanish version of the Mini-Mental State Examination. This is a 30-point questionnaire comprised by eight different categories and score range:
  Orientation to time (0-5 points) Orientation to place (0-5 points) Registration (0-3 points) Attention and calculation (0-5 points) Recall (0-3 points) Language (0-2 points) Repetition (0-1 points) Complex commands (0-6 points)
  The total score is the result of the summation of the categories. Interpretation:
  Any score greater than or equal to 24 points (out of 30) indicates a normal cognition.
  ≤9 points: severe cognitive impairment 10-18 points: moderate cognitive impairment 19-23 points: mild cognitive impairment
Assessment of the changes in participants' functional independence. | 10 weeks
  By means of the Barthel Index (BI) Spanish version. This scale evaluates the independence for the activities of daily living. It contains 10 different activities, with a possible score ranging from 0 to 10, with a maximum total score of the scale of 100 (summing the subscales results).
  Interpretation:
  <20 Total dependence 21 - 60 Severe dependence 61 - 90 Moderate dependence 91 - 99 Mild dependence 100 Total Independence
Assessment of the changes in participants' health-related self-perceived quality of life. | 10 weeks
  By means of the 12-Item Short-Form Health Survey (SF-12), spanish version. For each of the 8 subscales, the value can go from 0 to 100. For the interpretation of the results, the 50 (standard deviation 10) value on each dimension must be the mean valor for the sub scale reported for the general population, meaning that more or less than 50 must be considered better or worse, respectively.
Assessment of the changes in participants' fitness level. | 10 weeks
  By means of the 5-Chair Stands Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación San Rosendo, Panxón, Pontevedra, Spain